CLINICAL TRIAL: NCT05291650
Title: Ultrasound-guided Injection of Glucocorticoid Into Infrapatellar Fat Pad Versus Placebo Injection in Knee Osteoarthritis: a 12-week Double-blinded Controlled Trial
Brief Title: Ultrasound-guided Injection of Glucocorticoid Into Infrapatellar Fat Pad in Patients With Knee Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-KY-183-02
Record Dates: First submitted 2022-03-13; First posted 2022-03-23 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-09

CONDITIONS: Osteoarthritis, Knee
Keywords: knee osteoarthritis; infrapatellar fat pad; inflammatory osteoarthritis; glucocorticoid
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Glucocorticoids; Sodium Chloride; Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- glucocorticoid injection into infrapatellar fat pad (Active Comparator)
  Interventions: Drug: Glucocorticoids; Drug: Hyaluronic acid
- placebo injection into infrapatellar fat pad (Placebo Comparator)
  Interventions: Drug: Saline; Drug: Hyaluronic acid

INTERVENTIONS:
Drug: Glucocorticoids — The product of the glucocorticoid is betamethasone injectable suspension and the dosage is 1 ml. To alleviate the discomfort on local tissues, the suspension injected into the infrapatellar fat pad will be pre-mixed with 0.5 ml saline and 0.5 ml lidocaine. That is, the total amount of the drug injected into the infrapatellar fat pad for the glucocorticoid group will be 2.0 ml.
  Arms: glucocorticoid injection into infrapatellar fat pad
Drug: Saline — A total of 2.0 ml drug including 1.5 ml saline and 0.5 ml lidocaine will be injected into the infrapatellar fat pad for the placebo group.
  Arms: placebo injection into infrapatellar fat pad
Drug: Hyaluronic acid — After completing the process of infrapatellar fat pad injection, the participants in both groups will receive 2.5 ml hyaluronic acid suspension injection through the suprapatellar bursa into the intra-articular space.

SUMMARY:
This aims of this study is to investigate the efficacy and safety of the glucocorticoid injection into the infrapatellar fat pad among knee osteoarthritis patients with an inflammatory phenotype.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with symptomatic knee osteoarthritis (OA) according to American College of Rheumatology criteria;
2. Age > 45 years;
3. Have knee pain for more than six months and the knee pain over the past week assessed by VAS (100 mm) ≥ 40 mm;
4. Ultrasonography showed obvious synovitis with effusion in the knee joint;
5. Both MRI-assessed Hoffa-synovitis score (MOAKS method) and effusion-synovitis score (modified WORMS method) ≥ 1, and their total score ≥ 3;
6. Being able to listen, speak, read and understand Chinese, capable of understanding the study requirements and cooperating with the researchers during the study, and providing written informed consent.

Exclusion Criteria:

1. Allergy to glucocorticoids;
2. Knee injection of glucocorticoid or hyaluronic acid within the past six months;
3. Severe trauma or arthroscopy in the knee within the past six months;
4. Planned hip or knee surgery (including arthroscopy, arthroplasty, and other open joint surgeries) in the next six months;
5. Contraindication to having magnetic resonance imaging (MRI) (e.g., implanted pacemaker, artificial metal valve or cornea, aneurysm clipping surgery, arterial dissection, metal foreign bodies in the eyeball, claustrophobia);
6. Presence of other arthritis, such as rheumatoid arthritis and psoriatic arthritis;
7. Other physical condition that is more painful than their knee OA;
8. Malignant tumors or other life-threatening diseases;
9. Infection, diabetes, coagulopathy, osteonecrosis, or gastric/duodenal ulcer within the past 12 months;
10. Current use of oral corticosteroids, nonsteroidal anti-inflammatory drugs, or immunosuppressive medication;
11. Pregnancy or lactating female;
12. Use any investigational drugs or devices in the recent 30 days.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-12-26 (Actual)

PRIMARY OUTCOMES:
the knee pain change | over 12 weeks (assessed at baseline, the 4th week, the 8th week, and the 12th week)
  the knee pain change measured with visual analogue scale (VAS, 0-100), a higher VAS score means more severe pain
the change of effusion-synovitis volume | over 12 weeks (assessed at baseline and the 12th week)
  the change of magnetic resonance imaging assessed effusion-synovitis volume

SECONDARY OUTCOMES:
the change in WOMAC score | over 12 weeks (assessed at baseline, the 4th week, the 8th week, and the 12th week)
  WOMAC is an abbreviation for Western Ontario and McMaster Universities Osteoarthritis Index. WOMAC evaluates patients' pain (five items), stiffness (two items), and functional dysfunction (17 items) over the last week, with each item measured on a 100-mm visual analog scale. The WOMAC score is calculated by summing the scores of each item, with a higher WOMAC score indicating more severe OA symptoms.
the change in Hoffa-synovitis score | over 12 weeks (assessed at baseline and the 12th week)
  the Hoffa-synovitis score is assessed using the MRI Osteoarthritis Knee Score (MOAKS) method in MRI.
the change in quality of life | over 12 weeks (assessed at baseline, the 4th week, the 8th week, and the 12th week)
  quality of life is assessed using the four-dimensional Assessment of Quality of Life (AQoL-4D) questionnaire.
the change in pain medication use | over 12 weeks (assessed at baseline, the 4th week, the 8th week, and the 12th week)
  pain medication use is determined by the researchers from the records of medication use and categorized as commenced/increased, unchanged, or discontinued/decreased.
the change in Infrapatellar fat pad volume | over 12 weeks (assessed at baseline and the 12th week)
  the infrapatellar fat pad volume is assessed using MRI.
adverse reaction | the 4th week, the 8th week, and the 12th week
  adverse reactions are recorded at each follow-up, and the number of participants experiencing at least one adverse reaction is reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital, Guangzhou, China

REFERENCES:
- [Derived] Zhang Y, Ruan G, Fan T, Zheng P, Zhu Z, He J, Wei X, Hu W, Huang S, Chang Q, Gao P, Chen H, Zhou X, Liu X, Tang S, Jiang L, Ding C. Infrapatellar Fat Pad Glucocorticoid Injection in Knee Osteoarthritis: A Randomized Clinical Trial. JAMA Netw Open. 2026 Jan 2;9(1):e2549938. doi: 10.1001/jamanetworkopen.2025.49938. PMID 41481293
- [Derived] Zhang Y, Ruan G, Zheng P, Huang S, Zhou X, Liu X, Hu W, Feng H, Lin Y, He J, Wei Z, Zhang J, Chang Q, Wei X, Fan T, Jiang L, Ding C. Efficacy and safety of GLucocorticoid injections into InfrapaTellar faT pad in patients with knee ostEoarthRitiS: protocol for the GLITTERS randomized controlled trial. Trials. 2023 Jan 3;24(1):6. doi: 10.1186/s13063-022-06993-4. PMID 36597103